CLINICAL TRIAL: NCT02039232
Title: CarboFix Pedicle Screw System
Brief Title: Safety and Efficacy of the CarboFix Pedicle Screw System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CarboFix Orthopedics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARBOFIX P CLD PPS1
Record Dates: First submitted 2014-01-14; First posted 2014-01-17 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2018-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spinal Stenosis; Spinal Curvatures; Tumor
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spinal Stenosis; Spinal Curvatures; Neoplasms

ARMS (1):
- CarboFix Pedicle Screw System (Experimental)
  Interventions: Device: Pedicle screw system

INTERVENTIONS:
Device: Pedicle screw system

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CarboFix' Pedicle Screw System in the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years old or older.
2. Confirmation that the physical examination of radiopathy, myelopathy or combination is in correlation with the affected level.
3. Lumbar CT, MRI, or myelography confirms the level of involvement is consistent with the subject's examination.
4. Informed consent given by the subject.

Exclusion Criteria:

1. Subject is not eligible for fixation with market-available fixation means.
2. Familial history NF2.
3. Acute traumatic spinal injury with or without neurological signs.
4. Metabolic bone disease.
5. History of Paget's disease or other osteodystrophies whether acquired or congenital, including renal osteodystrophy, hyperthyroidism, hypothyroidism hyperparathyroidism, Ehrlers-Danlos-syndrome, osteogenesis imperfecta, achondroplasia, tuberculosis.
6. History of mental disorder or current psychiatric treatment.
7. Pregnancy and/or female subjects intending to become pregnant within the expected time frame of the study and/or female subjects of child bearing age who do not use conventional contraceptive methods.
8. Immune deficiency disease.
9. Infection in the location of the operative site, discitis, osteomyelitis, fever and/or leukocytosis (as diagnosed based on the results of CBC and ESR tests).
10. Scoliosis.
11. Treatment with drugs that may interfere with bone metabolism such as:

    1. Cumulative dose of 150 mg. of Prednisone or equivalent within the last 6 months.
    2. Calcitonin within the past 6 months.
    3. Bisphosphonates for 30 days or more within the last 12 months.
    4. Bone therapeutic doses of fluoride for 30 days or more within the last 12 months.
    5. Bone therapeutic doses of vitamin D or Vitamin D metabolites for 30 days or more within the last 6 months.
    6. Treatment by chemotherapy within the last 12 months.
12. Lack of willingness to make a commitment to return for required follow up visits.
13. Drug and/or alcohol abuse.
14. Morbid obesity.
15. Metal allergies.
16. Recent use of other investigational drugs or devices (within the past 30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Fusion success | 6 months post-operation

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hillel Yafe MC;, Hadera
  - Herzliya Medical Center, Herzliya